CLINICAL TRIAL: NCT03409250
Title: SD-OCT-guided Intravitreal Ranibizumab Treatment in Choroidal Neovascularization Due to Myopia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vista Klinik (Other)
Responsible Party: Principal Investigator, Dr. med. Katja Hatz, Dr. med. Katja Hatz, Vista Klinik
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MYOPIE-2011-04
Record Dates: First submitted 2014-11-25; First posted 2018-01-24 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Choroidal Neovascularization; Age Related Macular Degeneration
Keywords: CNV due to Age Related Macular Degeneration
MeSH Terms: conditions — Choroidal Neovascularization; Macular Degeneration | interventions — Ranibizumab; Intravitreal Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1-Arm study (Other): prospective, 1-arm, monocenter, investigator initiated study Intravitreal injection with Lucentis (Ranibizumab)
  Interventions: Drug: Ranibizumab, Lucentis

INTERVENTIONS:
Drug: Ranibizumab, Lucentis — Intravitreal injection with Lucentis (Ranibizumab)
  Other Names: Intravitreal injection with Lucentis (Ranibizumab)

SUMMARY:
This investigator initiated pilot study is designed to investigate the efficacy and safety of SD-OCT-guided intravitreal ranibizumab treatment in choroidal neovascularization (CNV) due to myopia. Newly diagnosed and active CNVs due to myopia are treated with one intravitreal injection of Ranibizumab 0.5mg (Lucentis) at baseline. During the follow up period of 12 months monthly ophthalmological examinations including best corrected visual acuity (BCVA) and high resolution spectral-domain optical coherence tomography (SD-OCT) assessments are performed. Detection of persisting or new signs of CNV activity at OCT triggers ranibizumab re-treatment considering that any ranibizumab injections can maximally be applied as often as monthly.

DETAILED DESCRIPTION:
Study purpose: This investigator iniiated pilot study is designed to investigate the efficacy and safety of SD-OCT-guided intravitreal ranibizumab treatment in choroidal neovascularization (CNV) due to myopia. Newly diagnosed and active CNVs due to myopia are treated with one intravitreal injection of Ranibizumab 0.5mg (Lucentis) at baseline. During the follow up period of 12 months monthly ophthalmological examinations including best corrected visual acuity (BCVA) and high resolution spectral-domain optical coherence tomography (SD-OCT) assessments are performed. Detection of persisting or new signs of CNV activity at OCT triggers ranibizumab re-treatment considering that any ranibizumab injections can maximally be applied as often as monthly.

Objectives: To investigate the efficacy and safety of SD-OCT-guided intravitreal ranibizumab treatment in choroidal neovascularization (CNV) due to myopia.

The primary objective is to demonstrate that a SD-OCT-guided intravitreal ranibizumab treatment in CNV due to myopia may prevent vision loss as evaluated as change in BCVA from baseline.

The secondary objectives are:

* To evaluate the changes in BCVA at 6 and 12 months compared to baseline.
* To evaluate the number of treatments needed at 6 and 12 months and the time course of re-treatments.
* To evaluate the time course of re-activation of CNV as evaluated by High Resolution OCT.
* To evaluate the incidence of fluorescein leakage as well as the mean and percent change in total area of CNV, total area of leakage from CNV, and total lesion area at 6 and 12 months.
* To evaluate the safety and tolerability of up to monthly dosing of ranibizumab in CNV due to myopia by determining the rates of adverse events and serious adverse events at month 6 and 12.

Population: This outpatient study population will consist of a representative group of male and female patients ≥ 18 years of age. The study population will include patients with newly diagnosed and active choroidal neovascularization (CNV) due to myopia. 20 Patients will be enrolled in one study center (Vista Klinik, Binningen).

Investigational and reference therapy:

This study will include the following study drug:

• Ranibizumab (Lucentis®) 0.5 mg for intravitreal injection.

Study design: This is a prospective, 1-arm, monocenter, investigator initiated study designed to evaluate the efficacy and safety of SD-OCT-guided intravitreal ranibizumab treatment in choroidal neovascularization (CNV) due to myopia. Newly diagnosed and active CNVs due to myopia are treated with one intravitreal injection of ranibizumab 0.5mg at baseline. During the follow up period of 12 months monthly ophthalmological examinations including best corrected visual acuity (BCVA) and high resolution spectral domain optical coherence tomography (SD-OCT) assessments are performed. Detection of persisting or new signs of CNV activity at OCT, as defined by intraretinal cysts or subretinal fluid, triggers ranibizumab re-treatment considering that any ranibizumab injections can maximally be applied as often as monthly.

For this study, a month is defined as 28 days. During the 12-month study period, a maximum of 12 ranibizumab injections may be administered.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age.
* Patients with active primary sub- or juxtafoveal CNV secondary to myopia.
* Evidence that CNV extends under the geometric center of the foveal avascular zone or in case of juxtafoveal lesions there is evidence that leakage from CNV extends under the geometric center of the foveal avascular zone as proven by fluorescein angiography.
* The total area of CNV encompassed within the lesion must be ≥ 50% of the total lesion area.
* The total lesion area ≤ 12 disc areas for minimally classic or occult with no classic component and ≤ 9 disc areas (5400µm) in greatest linear dimension with predominantly classic lesions.
* Patients who have a BCVA of ≥ 20/200 (letter score of ≥ 23 letters) in the study eye using ETDRS charts.
* Willing and able to give written informed consent according to legal requirements, and who have signed the consent form prior to initiation of any study procedure including withdrawal from exclusionary medications for the purpose of this study.
* Willing and able to comply with study procedures.

Exclusion Criteria:

* Subretinal hemorrhage in the study eye that involves the center of the fovea, if the size of the hemorrhage is either ≥ 50% of the total lesion area or ≥ 1 disc area in size.
* Structural damage to the center of the macula (beside CNV) in the study eye likely to preclude improvement in visual acuity, including atrophy of the retinal pigment epithelium, subretinal fibrosis, laser scar(s), or organized hard exudate plaques.
* Presence of a retinal pigment epithelial tear involving the macula in the study eye.
* Concurrent disease in the study eye that could compromise visual acuity or require medical or surgical intervention during the 12-month study period.
* Vitreous hemorrhage or history of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye.
* Active intraocular inflammation (grade trace or above) in the study eye.
* Any active infection involving ocular adnexa including infectious conjunctivitis, keratitis, scleritis, endophthalmitis, as well as idiopathic or autoimmune-associated uveitis in either eye.
* History of uncontrolled glaucoma in the study eye (defined as intraocular pressure ≥ 25 mmHg despite treatment with anti-glaucoma medication).
* Aphakia with absence of the posterior capsule in the study eye.
* Any prior treatment in the study eye with verteporfin, external-beam radiation therapy, subfoveal focal laser photocoagulation, vitrectomy, transpupillary thermotherapy, intravitreally applied drugs.
* History of submacular surgery in the study eye, glaucoma filtration surgery, corneal transplant surgery.
* Extracapsular extraction of cataract with phacoemulsification within three months preceding Baseline, or a history of post-operative complications within the last 12 months preceding Baseline in the study eye (uveitis, cyclitis, etc.).
* Use of other investigational drugs at the time of baseline, or within 30 days or 5 half- lives of baseline, whichever is longer (excluding vitamins and minerals).
* Previous violation of the posterior capsule in the study eye unless it occurred as a result of YAG posterior capsulotomy in association with prior, posterior chamber intraocular lens implantation.
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk for treatment complications.
* History of Stroke.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (>5 mIU/ml).
* History of hypersensitivity or allergy to fluorescein.
* Inability to obtain OCTs, fundus photographs or fluorescein angiograms of sufficient quality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
BCVA | Baseline to 12-months
  SD-OCT-guided intavitreal ranibizumab treatment in CNV due to myopiea may prevent vision loss as evaluated as change in BCVA from Baseline.

SECONDARY OUTCOMES:
BCVA change from Baseline to month 12 | Baseline to month 12
  To evaluate the changes in BCVA at 6 and 12 months compared to baseline.
Treatments from Baseline to month 12 | Baseline to month 12
  To evaluate the number of treatments needed at 6 and 12 months and the time course of re-treatments.
OCT changes from Baseline to month 12 | Baseline to month 12
  To evaluate the time course of re-activation of CNV as evaluated by High Resolution OCT.
Fluo changes from Baseline to month 12 | Baseline to month 12
  To evaluate the incidence of fluorescein leakage as well as the mean and percent change in total area of CNV, total area of leakage from CNV, and total lesion area at 6 and 12 months.
Ranibizumab tolerability from Baseline to month 12 | Baseline to month 12
  To evaluate the safety and tolerability of up to monthly dosing of ranibizumab in CNV due to myopia by determining the rates of adverse events and serious adverse events at month 6 and 12.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Pruente, MD, Principal Investigator — Vista Klinik
Locations (1):
- Vista Klinik, Binningen, Basel-Landschaft, Switzerland